CLINICAL TRIAL: NCT03318302
Title: University of Haifa
Brief Title: Sleep and Exposure to Screens of Digital Media Devices in Israel
Status: Completed | Type: Observational
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Lilach Kemer, Chief Dr., Assuta Medical Center
Other Study IDs: 039/17
Record Dates: First submitted 2017-10-14; First posted 2017-10-23 (Actual); Last update posted 2017-10-23 (Actual); Status verified 2017-10

CONDITIONS: Sleep Disturbance; Attention Deficit
MeSH Terms: conditions — Parasomnias; Attention Deficit Disorder with Hyperactivity | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Survey of the adult population in Israel
  Other Names: Survey of the adult population in Israel

SUMMARY:
The aims of this survey are to assess the relationships between exposure to screens of digital media devices, sleep patterns, and daily function such as subjective sleepiness and attention abilities in adult Israel population

DETAILED DESCRIPTION:
Self-reporting questionnaires: demographic, general health, sleep patterns and difficulties, and prevalence and exposure patterns to digital media screens.

1. Demographic: the participants report their age, gender, family status, education, and employment status including shift work.
2. General health: The subjective general health evaluation was measured with the question "Please rate how do you assess your health condition?" on a 5-point Likert scale with numbers and a description: 1 = "not good," 2 = "fine," 3 = "good," 4 = "very good," and 5 = "excellent." the participants report chronic sickness, prescription and non-prescription medications, height and weight, visual and sight condition ("Do you wear glasses? Do you suffer from cataracts?"). The participants self reports their level of concentration in the morning ("Please rate your level of concentration in the morning.") on a 9-point Likert scale. All of the numbers have valid point values, but only the odd numbers have descriptions: 1 = "extremely poor concentration", 3 = "not able to concentrate," 5 = "neutral, neither unable to concentrate or concentrate," 7 = "able to concentrate," and 9 = "extremely good concentration."
3. Sleep: The Pittsburgh Sleep Quality Index (PSQI) was applied to evaluate sleep timing, sleep onset latency, sleep duration, sleep difficulties, and sleep quality. The PSQI is a self-reporting questionnaire that assesses sleep quality over a 1-month time interval. The PSQI consists of 19 individual items comprising seven components that produce one global score. The PSQI is a standardized sleep questionnaire for clinicians and researchers to use with ease and for multiple populations, used in many research and clinical settings to diagnose sleep disorders (Buyess et al., 1989; Shocat et al., 2007). The Karolinska Sleepiness Scale (KSS) was used to assess sleepiness and tiredness. It is a nine-point Likert scale; all of the numbers have valid point values, but only the odd numbers have descriptions: 1 = "extremely alert," 3 = "alert," 5 = "neither alert nor sleepy," 7 = "sleepy," and 9 = "extremely sleepy" (Akerstedt and Gillberg, 1990; Gillberg et al., 1994)
4. Exposure to screens of digital media devices: The participants were asked about the presence and usage habits of digital media devices equipped with a screen (for example, TV, computer, tablet, and smartphone) and reported whether they had a TV, computer, tablet, and smartphone in their homes and bedrooms. They reported the duration of exposure time to digital screens of any digital media device for different time-periods of the day beginning in the morning until bedtime or sleep during weekdays and on weekends. We asked the participants to report on their exposure time to screens of digital devices the mean time in minutes of each separate time-period: early morning, before work or school, during work or study time, after work or study, until bedtime, and after bedtime. Digital media usage for all devices (TVs, computers, smartphones, and tablets) were computed for each 4-time periods of the day (sum-morning, Sum-day, sum-evening, and sum-night) reflecting the summation time in minutes to overall exposure time of digital media screens devices in each time segment of the day.

ELIGIBILITY:
Inclusion Criteria:

* All of the participants were Hebrew-speaking residents of Israel

Exclusion Criteria:

* under 18 years old No Hebrew-speaking residents of Israel

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult population of Isrel
Sampling Method: Probability Sample
Enrollment: 282 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
sleep quality | 30 days
  score on the PSQI questionnaire
subjective sleepiness | 30 days
  score on the KSS questionnaire
subjective concentration score | 30 days
  score on the concentration questionnaire
exposure time to digital screen | 30 days
  The exposure time to digital screens in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Lilach Kemer, Dr., Principal Investigator — Assuta Medial Center
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No